CLINICAL TRIAL: NCT02424825
Title: A Low-fat, Plant-based Cooking Course for Patients With Multiple Sclerosis
Brief Title: Rouxbe Pilot for MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Rouxbe Cooking School (Unknown)
Responsible Party: Principal Investigator, Vijayshree Yadav, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00011383
Record Dates: First submitted 2015-02-09; First posted 2015-04-23 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: diet; cooking; multiple sclerosis; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rouxbe (Experimental): Subjects will attend a one-month online cooking course, and be followed before, during, and after their participation for quality-of-life, fatigue, and blood biomarker changes.
  Interventions: Behavioral: Cooking Course

INTERVENTIONS:
Behavioral: Cooking Course — This is a month-long online cooking course, aimed at promoting a low-fat, plant-based diet.

SUMMARY:
The purpose of this protocol is to collect data from approximately 15 multiple sclerosis (MS) patients who are participating in a pilot cooking course. This online cooking training program is currently available to general public through the company "Rouxbe" for a fee. Data gathered from this cooking course will be used to develop novel ways of promoting healthy eating habits in people with MS. The investigators will use the data from blood tests, questionnaires, and demographics to assess the feasibility and effectiveness of this program. This is an outpatient program designed for people with MS that would occur regardless of whether participant data is collected.

This pilot cooking course will run for approximately four weeks. The investigators intend start to the training course in mid-March 2015. Subjects will be followed prior to course initiation for baseline data gathering, at four weeks from baseline, twelve weeks from baseline, and twenty-four weeks from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MS
* Willingness to comply with the diet and values set forth in the course

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Program Feasibility and Efficacy (composite of student perception, learning, and adherence by surveys) | 6 months
  We will measure feasibility as a composite of student perception, learning, and adherence by administering Opening and Closing Surveys (to evaluate student perception of course), a Final Assessment (to evaluate student learning), and the NutritionQuest Block Food Frequency Questionnaire (to evaluate adherence to low-fat, plant-based lifestyle).

SECONDARY OUTCOMES:
Weight Change measured by body weight, body mass index, waist circumference | 6 months
Diet Change measured by NutritionQuest Block Food Frequency Questionnaire, Opening Survey, Program Evaluation Survey | 6 months
Program Evaluation through Program Evaluation Survey | 6 months
Fatigue measured by Modified Fatigue Impact Scale-5 and Fatigue Severity Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vijayshree Yadav, MBBs, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University Multiple Sclerosis Center., Portland, Oregon, United States

REFERENCES:
- [Derived] Perlman J, Wu H, Fryman A, Lane M, Bittner F, Sammi MK, Rooney WD, Stevens A, Yadav V. Effects of vascular disease risk factors on brain metabolism in multiple sclerosis. Mult Scler Relat Disord. 2025 Dec;104:106700. doi: 10.1016/j.msard.2025.106700. Epub 2025 Sep 10. PMID 40976206
- See also: Rouxbe Cooking School — http://rouxbe.com/